CLINICAL TRIAL: NCT06071000
Title: Effect of Neurodevelopmental Stimulation on Motor and Cognitive Development in Neurotypical Healthy Children
Brief Title: Preschool Children Motor Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Motor development - Adam
Record Dates: First submitted 2023-07-21; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-01

CONDITIONS: Persisting Primitive Reflexes
Keywords: motor development; fundamental motor skills; executive functions; neurodevelopmental

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Behavioral: Neuro-developmental stimulation (Neuro-vývojová stimulace).
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Neuro-developmental stimulation (Neuro-vývojová stimulace). — Neuro-developmental stimulation is exercise based intervention program that is focused on repeating reflex movements and thus inhibiting reflexive response.
  Arms: Experimental group

SUMMARY:
The preschool age period is crucial for motor and cognitive development, which retention primary reflexes can negatively influence. Primary reflexes are fixed motor patterns controlled from developmentally lower areas of CNS and are necessary for delivery, survival or rudimentary movement activation during infancy and should be progressively inhibited. Primary reflexes' retention increases the risk of blocks for further cognitive and motor development in higher, mainly cortical areas. Children in preschool and school age with non-inhibited primary reflexes displayed a poor level of fundamental movement skills and worse attention, self-regulation or working memory capacity. Children with the problems above usually pass a movement program based on developmental kinesiology, like Neurodevelopmental stimulation (NVS). NVS contains exercises that simulate situations for adequate processing of the primary reflex and allow the brain to correct and inhibit this reflex. Even though in the Czech preschool environment, almost 13% of children with neurotypical development have significant positive responses to at least one primary reflex, there are no methods to inhibit primary reflexes to improve motor and cognitive development positively. Therefore, this project aims to find how the NVS intervention will influence the performance in the selected area of motor and cognitive development, with the follow-up three-month retesting. Population for this project are preschool children aged 4-6 years old.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* strong ADHD/learning disorders diagnosed

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
TGMD-2 | 8 months
  Test of gross motor development
IDS / IDS-P | 8 months
  Intelligence and Development Scale (preschool)
Primitive (primary) reflexes | 8 months
  Tests for persisting (retained) primitive reflexes